CLINICAL TRIAL: NCT06939192
Title: E-health-supported Recording of Psychological and Somatic Problems, Risk and Resilience Factors of Premature Born Infants and Their Families and Individualized, Interdisciplinary Stepped-care Approach
Brief Title: E-health-supported Diagnostic and Intervention in Preterm Born Children and Their Families
Acronym: NeoUp2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, PD Dr. Annette Conzelmann, Prof. Dr. Annette Conzelmann, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 652/2023BO2
Record Dates: First submitted 2025-03-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Preterm Birth
Keywords: Preterm birth; E-health; Risk factors; Protective factors; Prevention
MeSH Terms: conditions — Premature Birth | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (APP) (Experimental): The participants in the intervention group will be equipped with an app after inclusion in the study. The app contains specific information for parents with premature babies, a contact form for experts and questions about the child's development every 14 days.
  Interventions: Other: Intervention Group (APP)
- Treatment as usual Group (TAU) (Active Comparator): Participants in the treatment as usual group do not receive an app after inclusion in the study. They can contact their pediatrician if they have any questions.
  Interventions: Other: Treatment as usual-Group (TAU)

INTERVENTIONS:
Other: Intervention Group (APP) — Combination of app-based information and diagnostic screening for parents of premature babies.
  Arms: Intervention Group (APP)
Other: Treatment as usual-Group (TAU) — No intervention. Treatment in the form of usual aftercare service is possible.
  Arms: Treatment as usual Group (TAU)

SUMMARY:
The app-based diagnostic and support approach with a focus on mental and somatic symptoms is intended to strengthen the resilience of premature born children and families and to identify risk and resilience factors.The overall objective of the study is to improve the post-inpatient care of families with premature born children. The procedure is evaluated by a two-arm design with an experimental group and a TAU group.

DETAILED DESCRIPTION:
The project aims to conduct a longitudinal study of premature babies and their parents from the time of hospital discharge in order to identify predictive factors for their psychological and physical outcomes and to provide individualized interdisciplinary diagnostic and treatment. The project helps to identify risk and protective factors and also takes a closer look at the interplay between the mind and body. This care approach is supported by an app that records symptoms and needs and also allows contact with the study team. The app also provides psychoeducational materials. The study was developed in collaboration with affected families and experts from the aftercare team. The concept will be evaluated by comparing the treatment group with a TAU group and by conducting measurements after hospital discharge, after 4 months, and again after 7 months, as well as through focus groups with study participants.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies born at the UKT,
* Gestational age 28-34 weeks,
* Mother: age ≥ 18 years,
* agreement to participate in this study and signing of a consent form,
* sufficient knowledge of German,
* internet access

Exclusion Criteria:

* Premature babies < 28th or >34th week of pregnancy,
* at least one of the children has serious diseases of the nervous system or obvious symptoms of a nervous disease,
* at least one of the children has serious congenital diseases or suffers from malformations,
* Mother: Lack of access to a smartphone/tablet,
* no internet access,
* insufficient knowledge of German

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on satisfaction, feasibility, needs (FB-NB) | At month 4 (post-teatment, T1) and month 7 (follow-up, T2)
  After completion of the main study phase, the self-constructed questionnaire assesses satisfaction with the study concept and evaluates the feasibility of the study approach. Patients are asked to indicate their satisfaction using a Likert scale and can also note down any additional or modification requests in free text fields.
Parent Stress Inventory (EBI) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The EBI measures the extent of parental stress and contains 48 items that are assigned to 12 subscales. Answering on a Likert scale.
Crying, Feeding and Sleeping Questionnaire (SFS) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The questionnaire on regulatory disorders in childhood uses 54 questions to assess early childhood regulatory disorders in relation to crying, eating or sleeping. The response format is generally a 4-point scale from not at all to very much.

SECONDARY OUTCOMES:
Demographic data | At baseline (before treatment, T0).
  The questionnaire includes, among other things, the age, gender, ethnicity and socio-demographic data of the test subjects.
Brief Symptom Inventory (BSI) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The questionnaire is a short form of the SCL-90-R and measures the subjectively perceived impairment of a person through physical and psychological symptoms on nine scales (somatization, compulsiveness, insecurity in social contact, depressiveness, anxiety, aggressiveness / hostility, phobic anxiety, paranoid thinking, psychoticism) with 53 items, within a period of 7 days. Answering the questions on a Likert scale from 0 to 4.
Brief Infant Sleep Questionnaire (BISQ) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The BISQ is a short and simple questionnaire about the child's sleep duration, nocturnal awakenings and methods of falling asleep.
Edinburgh Postnatal Depression Scale (EPDS) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The EPDS measures depression in the last 7 days with 10 items.
Couple Conflict Questionnaire (PFB-K) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The partnership questionnaire measures the quality of the partnership with only 9 items in 3 subcategories (argumentative behavior, tenderness, communication), answered on a Likert scale.
Parent-Child Relationship Questionnaire (PBQ) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The PBQ is an instrument for assessing the quality of the postpartum relationship between mother and child. The questionnaire comprises 25 items and is answered on a Likert scale from 1 to 6.
Ulm Quality of Life Inventory for Parents (ULQIE) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The questionnaire comprises a total of 29 items on the well-being and quality of life of the parent, covering a period of one week, answered on a five-point Likert scale from 0 (never) to 5 (always).
Ages & Stages Questionnaire®: Third Edition (ASQ-3) | At month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The questionnaire is a developmental screening tool that measures developmental progress in children aged 1 month to 5 ½ years. It comprises a total of 30 questions, 6 for each developmental area on child communication, fine and gross motor skills, problem solving and social behavior.
Focus groups | At baseline (before treatment, T0), after month 7 (follow-up, T1).
  Conducting several focus groups with parents and professionals on the needs of post-inpatient care for parents with a premature baby. Survey of needs and feedback from the app group.
App-questions | Every 14 days over a period of 4 months (baseline, T0 - post-treatment, T1).
  Questions about the child's and parents' state of health, well-being and perception of stress
Questionnaire on health economics (HCU-Q) | At month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  The translated questionnaire for measuring the use of healthcare services was developed based on the Health Care Utilization Questionnaire. Due to the young age of the children, some items were replaced. The questionnaire is intended to assess the families' respective use and utilization of medical and non-medical health care services.
Self-efficacy questionnaire (SWE) | At baseline (before treatment, T0), at month 4 (post-teatment, T1) and month 7 (follow-up, T2).
  10 items on dealing with difficult situations and one's own perceived self-efficacy, answered on a scale from 1 (not true) to 4 (true).

CONTACTS AND LOCATIONS:
Overall Officials: Annette Conzelmann, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University of Tübingen; Annika K Alt, Study Chair — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University of Tübingen; Tobias J Renner, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University of Tübingen; Axel Franz, Prof. Dr., Study Chair — Neonatology, University of Tübingen; Mirja Quante, Dr., Study Chair — Neonatology, University of Tübingen; Michaela Minarski, Dr., Study Chair — Neonatology, University of Tübingen; Johanna Löchner, Prof. Dr., Study Chair — Clinical Psychology, FAU Erlangen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
We share study material and statistical outputs.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Any time before and after completion of the study for 10 years.
Access Criteria: Upon request.